CLINICAL TRIAL: NCT03562624
Title: Multi-center, Randomized, Comparator-controlled, Single-blind, Parallel-Group Study to Investigate the Pharmacodynamics, Pharmacokinetics and Safety of an Intrauterine System (BAY987443) With Three Different Release Rates of Indomethacin and One Release Rate of Levonorgestrel, as Compared With Jaydess, in a Combined Proof-of-concept and Dose Finding Study in Healthy Pre-menopausal Women Treated for 90 Days
Brief Title: A Study to Compare 3 Doses of a Hormonal Intra-uterine Device Containing Levonorgestrel and Indomethacin With a Hormonal Intra-uterine Device Containing Only Levonorgestrel to Assess the Effect and Safety of the Combined Components
Acronym: INDessa
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17700; 2018-000128-33 (EudraCT Number)
Record Dates: First submitted 2018-06-08; First posted 2018-06-19 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-08

CONDITIONS: Contraception
MeSH Terms: interventions — Levonorgestrel

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BAY98-7443 (low IND dose) (Experimental): Combi IUS Treatment, LNG (Levonorgestrel) with lowest dose of IND (indomethacin)
  Interventions: Drug: BAY98-7443
- BAY98-7443 (middle IND dose) (Experimental): Combi IUS Treatment, LNG with medium dose of IND
  Interventions: Drug: BAY98-7443
- BAY98-7443 (high IND dose) (Experimental): Combi IUS Treatment, LNG with highest dose of IND
  Interventions: Drug: BAY98-7443
- Marketed comparator (Active Comparator): Marketed comparator IUS
  Interventions: Drug: Levonogestrel (Skyla, BAY86-5028)

INTERVENTIONS:
Drug: BAY98-7443 — Active ingredient content (in mg IND/LNG):
  low dose 6.5 / 13.5; middle dose 12.5 / 13.5; high dose 15.4 / 13.5
  Arms: BAY98-7443 (high IND dose); BAY98-7443 (low IND dose); BAY98-7443 (middle IND dose)
Drug: Levonogestrel (Skyla, BAY86-5028) — Comparative LNG dose
  Other Names: Jaydess
  Arms: Marketed comparator

SUMMARY:
This study is the first study investigating the combined intrauterine administration of LNG (levonorgestrel) and IND (indomethacin). It is a combined proof-of-concept (PoC) and dose finding (DF) study in pre-menopausal women. It is designed to investigate the pharmacodynamics (PD) of BAY 987443 (i.e. IUS (intrauterine system) releasing LNG and IND), as well as pharmacokinetics (PK) of both active substances, safety and tolerability. In this study, Jaydess, as an LNG-only IUS, will be used as a comparator.

ELIGIBILITY:
Inclusion Criteria:

* Agreement to use an acceptable non-hormonal method of contraception (i.e. male or female condom with or without spermicide; cap, diaphragm or sponge with spermicide) when sexually active. This applies during the pre-treatment cycle and directly following the treatment period until the end of the follow-up period. This is not required if safe contraception is achieved by a permanent method, such as bilateral fallopian tube blockage of the subject or vasectomy of the partner(s).
* Age at screening: 18-45 years inclusive
* Body mass index (BMI) at screening: ≥ 18 and ≤ 32 kg/m²
* No clinically relevant abnormal findings in the pre-treatment endometrial biopsy
* Adequate venous access (for frequent blood sampling)

Exclusion Criteria:

* Menstrual disorders with unknown reason (not e.g. oligomenorrhea, hypomenorrhea amenorrhea due to hormonal treatment; not irregularities occurring during menarche). In case it is suspected that the woman is peri-menopausal, she should be excluded.
* Use of short-acting hormonal contraceptives/preparations containing sex hormones (oral, transdermal, intravaginal, IUS) during the pretreatment cycle
* Use of long-acting preparations containing sex hormones within the 40 weeks before the first screening examination (any long-acting injectable or implant)
* History of known or presence of suspected or known malignant tumors, especially any breast cancer, cervical carcinoma in situ or other progestin-sensitive cancer
* History of skin reactions, or other allergic-type reactions or known hypersensitivity reactions after taking aspirin, IND or other NSAIDs or to LNG, or any excipients of the IUSs
* Regular use of corticosteroids, irrespective of route of administration
* Known asthma bronchiale and aspirin-sensitive asthma
* Current or recurrent pelvic inflammatory disease
* Abnormal cervical smear within the last 6 month prior to screening
* Acute genital infection
* Known current thyroid disorders which require treatment (subjects with an euthyroid struma who do not need any treatment can participate)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2018-06-22 (Actual); Primary Completion 2019-05-16 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Number of uterine bleeding/spotting (B/S) days during treatment | 90 days after start of treatment
  Recorded by participants with electronic diary

SECONDARY OUTCOMES:
Number of subjects showing endometrial histology typical for intrauterine LNG application in biopsies taken at the end of treatment | On day 90 after start of treatment
Frequency of treatment emergent adverse events | 90 days after start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (7):
- Germany (6):
  - Nuvisan GmbH, Neu-Ulm, Bavaria
  - Frauenarztpraxis Dr. Wetzel, Blankenburg, Saxony-Anhalt
  - Dinox GmbH Berlin, Berlin
  - CRS Clinical Research Services Berlin GmbH, Berlin
  - CTC North GmbH & Co. KG, Hamburg
  - Praxis Hr. Dr. K. Peters, Hamburg
- PAREXEL International Early Phase Clinical Unit (London), Harrow, United Kingdom

REFERENCES:
- [Derived] Hofmann BM, Ahola M, Fels LM, Klein S, Lindenthal B, Pihlaja J. Development of an Intrauterine Device Releasing Both Indomethacin and Levonorgestrel During the First Months of Use: Pharmacokinetic Characterization in Healthy Women. Clin Pharmacokinet. 2023 Jan;62(1):113-126. doi: 10.1007/s40262-022-01201-7. Epub 2023 Jan 17. PMID 36648744